CLINICAL TRIAL: NCT06413927
Title: A Contemporary Look at Driver Training and Its Role in Reducing Crash Risk in Novice Adolescent Drivers
Brief Title: Driver Education Research Study
Acronym: DRIVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Pennsylvania (Other); University of Michigan (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-019445; 1R01HD108249-01A1 (NIH)
Record Dates: First submitted 2024-04-24; First posted 2024-05-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Risk Reduction Behavior; Injuries; Accident, Traffic; Development, Adolescent
Keywords: Injury prevention; Adolescent development; Learner drivers; Crash risk reduction; Novice drivers; Risky Driving; Teens
MeSH Terms: conditions — Risk Reduction Behavior; Wounds and Injuries

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The research staff who are unblinded will deliver the electronic surveys and cognitive battery (which is automatically scored) at baseline before participants are randomly assigned to an arm. The primary outcome variables are automatically scored, thus blindly to intervention arm. The Virtual Driving Assessment is a self-guided tool and is automatically scored. The smartphone app automatically records hard braking events and other behaviors without knowledge of intervention arm. Licensing tests will be conducted by state-sanctioned licensing examiners who will be blinded to which arm the participant is in (per state mandate).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Control: Online Vehicle and Driver Safety Education (Active Comparator): Participants in this arm will receive care as usual, and also complete an online video training module on vehicle and driver safety, with a short quiz at the end to determine compliance. The training content will not teach driving skills, as in the other online driver training arm. It requires up to two hours to complete and can be done from any internet-connected computer (at home, at school, etc.).
  Interventions: Behavioral: Online Vehicle and Driver Safety Education
- Online Driver Skills Training (Experimental): Participants in the Online Driver Skills Training arm will complete an online driver skill training program known as Accelerated Curriculum to Create Effective Learning (ACCEL) for novice drivers. It requires up to two hours to complete and can be done from any internet-connected computer (at home, at school, etc.).
  Interventions: Behavioral: Online Driver Skills Training
- Behind-the-Wheel Driver Training (Experimental): Participants in the Behind-the-Wheel training arm will receive professional behind-the-wheel training course delivered in-person on the road by a local driving school instructor through our partnership with a local driving school Coastline Academy.
  Interventions: Behavioral: Behind-the-Wheel Driver Training

INTERVENTIONS:
Behavioral: Online Vehicle and Driver Safety Education — This online video education program provides education in vehicle and driver safety (e.g. vehicle maintenance, adjusting car seats and seatbelts). This online training will take up to 2 hours to complete and will have a short quiz at the end to determine compliance with this online training.
  Arms: Active Control: Online Vehicle and Driver Safety Education
Behavioral: Online Driver Skills Training — The online driver training is the Accelerated Curriculum to Create Effective Learning (ACCEL) is designed to enhance the ability to anticipate, recognize and respond to hazards and to maintain attention to the road. The training is delivered online via a computer and can be done from home or at a school or other site that has a computer with internet access. It requires up to two hours to complete, and will be hosted on a platform that will track progress and completion through the training (such as accuracy, duration in modules, time to complete) and a short quiz will be provided at the end to assess learning.
  Arms: Online Driver Skills Training
Behavioral: Behind-the-Wheel Driver Training — The professional behind-the-wheel training course will be conducted in-person, delivered by local driving school partner Coastline Academy. The curriculum consists of 6 hours of training with assigned practice between lessons, and meets Pennsylvania and national standards. Post-lesson forms completed by the instructors will record adherence and consistency (intervention fidelity).
  Arms: Behind-the-Wheel Driver Training

SUMMARY:
This study will test the effectiveness of different types of driver training interventions for reducing young new driver crash risk early after licensure.

DETAILED DESCRIPTION:
Motor vehicle crashes remain high in young drivers, despite graduated driver licensing laws that put restrictions on driving and delay licensure. Typically, data trends show that crash risk is highest right after licensure, in the early months of independent driving. Additional studies of different driver training interventions have shown some evidence that it is possible to improve skills and reduce crashes early in licensure for young drivers. However, Pennsylvania and many other states have no professional training requirements for young drivers.

This study will test the effectiveness of different types of driver training programs for reducing young new driver crash risk early after licensure.

Up to 1,200 adolescent learner drivers in Pennsylvania will be recruited for this trial (to get up to 1,000 evaluable participants). Participants will be recruited through Primary Care Clinics at Children's Hospital of Philadelphia and from the surrounding community to take part in a study that will continue through the learner phase and for 6 months after licensure. Participants will give informed consent and be asked to complete some baseline surveys and cognitive tasks, and a virtual driving assessment in-person during a clinical or other visit. All will receive care-as-usual.

Participants will also be followed through the learner phase with a smartphone app that monitors driving trips and monthly surveys that can be completed at home. In the learner phase, participants will randomly receive one of three interventions. One group of participants will receive professional behind-the-wheel training with a local driving school instructor. Another group will receive a modern online driver training course. Another group will receive an online vehicle and driver safety education. Participants randomly assigned to the behind-the-wheel training group will be required to download and use an app to log and track their driving practice hours. Use of this app will be optional for participants randomly assigned to the other groups.

After the learner phase, participants will be given an online hazard skills test, online surveys, and second virtual driving assessment, and state license examination and will be followed for 6 months after licensure, with online surveys at 2, 4, and 6 months after licensure, and with continued driver trip monitoring through the smartphone app.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 16-17 years old who reside in Pennsylvania
* Have an active Pennsylvania learner's permit
* Have <30 hours of driving practice during permit phase
* Have never taken an on-road licensing exam, in any state
* Plan to get a license within the next 12 months in Pennsylvania
* Plan to have access to a vehicle to drive after licensure
* Have a personal cell phone and access to a smartphone/tablet/computer with internet access
* Download and use the RoadReady app (only required for participants randomized to the behind-the-wheel training arm; optional for participants randomized to the online vehicle and driver safety and online driver skills training arms)
* Are able to read/write in English
* Provide informed consent/assent
* Are not also taking part in another learner driver study

Exclusion Criteria:

* Non-Pennsylvania resident
* Participants who do not pass the license exam will not be able to complete the post-license monitoring until the license is obtained
* Enrolled in another learner driver study

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1300 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Hard Braking Events | Measured over the 6 months post-licensure at the end of the study (about month 18-24), assessed at 2 and 6 months post-licensure, with primary outcome at 2 months post-licensure.
  For Aim 1 and 3, the primary outcome is the number of hard braking events per 100 miles driven during the first 2 months post-licensure, as measured via the Way-to-Drive App.
Pass rate on the licensure exam | Measured at the time of the license examination, post-intervention (in about month 8-18).
  The primary outcome in Aim 2 and 3 will be the pass rate on the first licensure exam attempt.

SECONDARY OUTCOMES:
Phone Use While Driving | Measured over the 6 months post-licensure at the end of the study (about month 18-24), assessed at 2 and 6 months post-licensure.
  For Aim 1 and 3: minutes of handheld phone use per hour of driving, as measured via the Way-to-Drive App.
Speeding | Measured over the 6 months post-licensure at the end of the study (about month 18-24), assessed at 2 and 6 months post-licensure.
  For Aim 1 and 3: Proportion of drive time >10 miles over the posted speed limit, as measured via the Way-to-Drive App.
Crash Involvement | Measured at 2-, 4- and 6-month follow-up post-licensure (about month 18-24).
  For Aim 1 and 3: Self-reported involvement in crashes as a driver (binary yes/no) as captured by a question in our follow-up driver experience questionnaire: response options are 1) none; 2) one; 3) two; 4) more than 2. This item has been used in previous studies as part of the modified Driver Behavior Questionnaire (mDBQ).
Risky driving behavior | Measured at 2-, 4- and 6-month follow-up post-licensure (within about month 18-24).
  For Aim 1 and 3: Risky Driving factor score as captured through self-reported responses on the modified driver behavior questionnaire, in which participants rate how often they engage in 11 different risk-taking behaviors while driving on a 6-point scale from "Never" to "Nearly all the time."
Virtual Driving Assessment performance | Measured at the time of the license examination, post-intervention (in about month 8-18).
  For Aim 2 and 3: the class of driving behavior assessed via performance on a virtual driving assessment.
Change in Virtual Driving Assessment performance | Measured at the time of the license examination, post-intervention (in about month 8-18).
  For Aim 2 and 3: the change in virtual driving assessment performance class assessed via performance on a virtual driving assessment pre- and post-intervention.
Number of license exam attempts | Measured at the time of the license examination, post-intervention (in about month 8-18).
  For Aim 2 and 3: the number of attempts taken to pass the licensure exam.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Walshe, PhD, Principal Investigator — Children's Hospital of Philadelphia; Flaura Winston, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia; Dan Romer, PhD, Principal Investigator — Children's Hospital of Philadelphia/University of Pennsylvania
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walshe EA, Romer D, Elliott MR, Baxelbaum KS, Delgado MK, Ebert JP, Winston FK. A contemporary examination of the effect of driver training for reducing crash risk in novice adolescent drivers: protocol for the DRIVER study, a random assignment trial. Inj Epidemiol. 2025 Dec 1;13(1):2. doi: 10.1186/s40621-025-00645-2. PMID 41327408